CLINICAL TRIAL: NCT02735863
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase IIa Trial to Compare the Safety of ABX464 Given at a Fixed Dose to Placebo in Fully Controlled HIV Infected Patients Treated With Boosted Protease Inhibitor Treatment (Darunavir/Ritonavir or Darunavir/Cobicistat).
Brief Title: ABX464 in Fully Controlled HIV Infected Patients Treated With Boosted Protease Inhibitor Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-004
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-06

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — ABX464

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABX464 (Experimental): Fixed dose of ABX464 50mg once daily given during 28 days in association with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI)
  Interventions: Drug: ABX464
- ABX464 Matching placebo (Placebo Comparator): Matching placebo of ABX464 given at 50mg once daily in association with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — 50 mg or 150mg once daily for 28 days
  Arms: ABX464
Drug: Placebo — ABX464 matching placebo
  Arms: ABX464 Matching placebo

SUMMARY:
This study is a placebo-controlled study aimed at assessing the safety of ABX464 administered at 50 mg and 150 mg o.d. versus placebo in HIV infected patients who are treated with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI).

DETAILED DESCRIPTION:
This study is a placebo-controlled study aimed at assessing the safety of ABX464 administered at 50 mg o.d. and 150 mg versus placebo in HIV infected patients who are treated with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI). Eligible patients should be treated with darunavir + ritonavir or darunavir + cobicistat as monotherapy for at least 8 weeks prior to baseline. Patients should be fully suppressed (< 50 copies/mL) at least during the last 6 months prior to enrolment.

Upon screening visit, eligible patients will continue DRV/RTV or DRV/COBI single regimen given respectively at 800 mg of darunavir with 100 mg of ritonavir or 150 mg of cobicistat once a day with food in the morning.

At Day 0, study drug (ABX464 or its matching placebo) will be added on top of this background therapy for the next 28 days. ABX464 or its matching placebo will be given once a day at 50 mg or 150 mg.

At day 29, DRV/RTV or DRV/COBI and ABX464 or its matching placebo (i.e. all treatments) will be stopped. The viral load will be monitored twice a week during the first three weeks and weekly during the next weeks. In case of Viral Rebound (VR; defined below), ART will be resumed.

A 3:1 randomization ratio will be applied meaning that, per treatment block, 3 patients will receive ABX464 on top of DRV/RTV or DRV/COBI and 1 patient will receive placebo on top of DRV/RTV or DRV/COBI.

Dose limiting toxicity (DLT) is defined as a grade 3 or higher adverse event as defined by the "Division of AIDS table for grading the severity of adult and pediatric adverse events" (including signs/symptoms, lab toxicities and/or clinical events) considered by the Data Safety Monitoring Board as probably or definitely related to study treatment.

If more than 2 DLTs occur during the treatment period of the first four treated patients, then the enrolment of additional patients will be stopped. In addition, in case of a life threatening (grade 4) adverse reaction enrolment and treatment of ongoing patients will be immediately discontinued. In both cases, enrolment will only be resumed upon the decision of the sponsor if the Data Safety Monitoring Board can conclude that the causality of the event was unrelated or unlikely related to study treatment.

Thorough pharmacokinetics analysis will be performed to characterize potential drug-drug interactions between ABX464 and DRV/RTV-COBI.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with HIV;
* Patients with HIV plasma viral load ≤ 50 copies mL-1 during the 6 months prior to screening with a maximum of 2 blips during this period;
* Patients treated by DRV/RTV or DRV/COBI as a monotherapy for at least 8 weeks prior to baseline;
* Patients' HIV plasma viral load ≤100,000 copies mL-1 at any time (apart from primary infection if recorded);
* Patients' CD4+ T cells count ≥ 250 cells per mm3 at any time since diagnosis;
* Patients with CD4+ T cells count ≥ 600 cells per mm3 at screening;
* Man or woman aged 18-65 years;

Exclusion Criteria:

* Patient displaying any HIV protease inhibitor resistance mutation as listed in the current version of the HIV drug resistance database (Stanford University);
* Patient having had previously a viral load ≥ 500 copies mL-1 confirmed by a second measure since the initiation of the current ART;
* History of an AIDS-defining clinical illness;
* Concomitant AIDS-related opportunistic infection;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08-30 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (3):
  - C.H.U. Saint-Pierre, Brussels
  - Ghent University Hospital, Ghent
  - CHU Sart Tilman, Liège
- France (2):
  - Hôpital de la Croix Rousse, Lyon
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
- Spain (3):
  - Hospital Clinic, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari Germans Trias i Pujo, Barcelona

REFERENCES:
- [Derived] Rutsaert S, Steens JM, Gineste P, Cole B, Kint S, Barrett PN, Tazi J, Scherrer D, Ehrlich HJ, Vandekerckhove L. Safety, tolerability and impact on viral reservoirs of the addition to antiretroviral therapy of ABX464, an investigational antiviral drug, in individuals living with HIV-1: a Phase IIa randomised controlled study. J Virus Erad. 2019 Jan 1;5(1):10-22. doi: 10.1016/S2055-6640(20)30273-9. PMID 30800421

RESULTS

PARTICIPANT FLOW:
Groups:
- ABX464 50mg: Fixed dose of ABX464 50mg once daily given during 28 days in association with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI)
- ABX464 150mg: Fixed dose of ABX464 150mg once daily given during 28 days in association with darunavir + ritonavir (DRV/RTV) or darunavir + cobicistat (DRV/COBI)
Period: Overall Study
Arm/Group | ABX464 50mg | ABX464 150mg | ABX464 Matching Placebo
Started | 6 | 16 | 8
Completed | 5 | 14 | 7
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Patients who had received at least one dose of the study drug, and who had at least one baseline value.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABX464 50mg | ABX464 150mg | ABX464 Matching Placebo | Total
Number analyzed (Participants) | 6 | 16 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 16 | 8 | 30
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (3.5) | 38.4 (10.4) | 48.3 (8.5) | 42.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 6 | 15 | 8 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 6 | 14 | 7 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 10 | 4 | 17
  France | 0 | 1 | 1 | 2
  Spain | 3 | 5 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Patients who had received at least one dose of the study drug, and who had at least one baseline value. An AE was classified as a TEAE if it started, or increased in severity, on or after the first date and time of medication dosing (from Day 1 up to Day 28). Any AE which occurred after Day 28 was classified as post-treatment-emergent. Events were graded according to the "Division of AIDS table for grading the severity of adult and pediatric adverse events" (Version 2.0 November 2014).
Time Frame: Up to 4 months
Population: Patients who had received at least one dose of the study drug, and who had at least one baseline value.
Measure: Count of Participants; unit: Participants
Arm/Group | ABX464 50mg | ABX464 150mg | ABX464 Matching Placebo
Number analyzed (Participants) | 6 | 16 | 8
Participants
  Any AE | 5 | 15 | 7
  Any TEAE | 4 | 15 | 3
  Any post-TEAE | 4 | 6 | 4
  Any serious AE | 0 | 0 | 1
  Any severe AE | 0 | 1 | 0
  AE leading to death | 0 | 0 | 0

2. Secondary Outcome: Time to Viral Rebound
Description: Time To Viral Rebound is defined as the time between treatment stop (i.e. day 29) and viral rebound detection
Time Frame: Up to 3 months
Population: Patients who had received at least one dose of the study drug, and who had at least one baseline value.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABX464 50mg | ABX464 150mg | ABX464 Matching Placebo
Number analyzed (Participants) | 6 | 16 | 8
days | 17.2 (3.4) | 14.4 (7.4) | 14.4 (7.3)
Statistical Analysis 1: Comparison: ABX464 50mg vs ABX464 150mg vs ABX464 Matching Placebo; Test type: Superiority; p = 0.5352, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 4 months
Description: Patients who had received at least one dose of the study drug, and who had at least one baseline value.
Arm/Group | ABX464 50mg | ABX464 150mg | ABX464 Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/16 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/16 | 1/8
Other Adverse Events (participants affected / at risk) | 5/6 | 15/16 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg (N=6) | ABX464 150mg (N=16) | ABX464 Matching Placebo (N=8)
vagal faintness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABX464 50mg (N=6) | ABX464 150mg (N=16) | ABX464 Matching Placebo (N=8)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (5) | 0 (0)
Influenza Like Illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
C-reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (7) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02735863/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02735863/SAP_001.pdf